CLINICAL TRIAL: NCT04962815
Title: Ceribell Delirium Data Collection Study
Status: Recruiting | Type: Observational
Sponsor: Ceribell Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2021-01
Record Dates: First submitted 2021-06-29; First posted 2021-07-15 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Delirium
Keywords: delirium; EEG; Electroencephalogram
MeSH Terms: conditions — Delirium | interventions — Electroencephalography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Electroencephalogram (EEG) Test — EEG test and delirium assessments will be performed on subjects experiencing delirium in the ICU.
  Other Names: Delirium Assessments

SUMMARY:
This study is designed as a prospective, non-randomized, observational clinical study. The study will collect clinical and rrEEG (Ceribell EEG) data when monitoring subjects for delirium subtypes. EEG and clinical data will be collected for the development of future software algorithms to assess the presence and severity of delirium.

ELIGIBILITY:
Inclusion Criteria: All must be present

* Age is 18 years or older
* Admitted to the Intensive Care Unit (ICU)
* Subject must be fluent in the language in which the delirium assessment is performed

Exclusion Criteria: All must be absent

- Any condition that prevents use of the Ceribell EEG system on the subject for the entire anticipated EEG monitoring period. Examples may include: Craniectomy with missing bone flap in an area where Ceribell EEG electrodes are placed. Expected use of continuous clinical EEG for the entire anticipated monitoring period.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects who experience at least one delirious episode during their ICU stay
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-11-10 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Perform Confusion Assessment Method for the ICU (CAM-ICU) assessment | 3 times per day, for a maximum of six (6) days
  Research coordinator will perform and collect CAM-ICU assessment data on study subjects
Perform Electroencephalogram (EEG) Test | 6-8 hours per day, for a maximum of six (6) days
  Record and collect EEG brain waves on study subjects using Ceribell Rapid Response EEG to assess multiple time-frequency EEG features to differentiate between delirium positive and delirium negative patients.

CONTACTS AND LOCATIONS:
Overall Officials: Jose Maldonado, MD, Principal Investigator — Stanford University; Timothy Girard, MD, Principal Investigator — University of Pittsburgh
Locations (7):
- United States (7):
  - Stanford University, Stanford, California
  - Naples Community Hospital, Naples, Florida
  - University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - Mercy, St Louis, Missouri
  - Cooper Health, Camden, New Jersey
  - UNC Health Rex, Raleigh, North Carolina
  - University of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Site investigators will have access to the participant EEG data via Ceribell EEG portal. In addition, site investigators will have access to delirium assessments conducted for study purposes.
Supporting Information: Study Protocol, ICF

REFERENCES:
- [Background] Ely EW, Shintani A, Truman B, Speroff T, Gordon SM, Harrell FE Jr, Inouye SK, Bernard GR, Dittus RS. Delirium as a predictor of mortality in mechanically ventilated patients in the intensive care unit. JAMA. 2004 Apr 14;291(14):1753-62. doi: 10.1001/jama.291.14.1753. PMID 15082703
- [Background] Pandharipande P, Cotton BA, Shintani A, Thompson J, Pun BT, Morris JA Jr, Dittus R, Ely EW. Prevalence and risk factors for development of delirium in surgical and trauma intensive care unit patients. J Trauma. 2008 Jul;65(1):34-41. doi: 10.1097/TA.0b013e31814b2c4d. PMID 18580517
- [Background] McPherson JA, Wagner CE, Boehm LM, Hall JD, Johnson DC, Miller LR, Burns KM, Thompson JL, Shintani AK, Ely EW, Pandharipande PP. Delirium in the cardiovascular ICU: exploring modifiable risk factors. Crit Care Med. 2013 Feb;41(2):405-13. doi: 10.1097/CCM.0b013e31826ab49b. PMID 23263581
- [Background] Maldonado JR. Acute Brain Failure: Pathophysiology, Diagnosis, Management, and Sequelae of Delirium. Crit Care Clin. 2017 Jul;33(3):461-519. doi: 10.1016/j.ccc.2017.03.013. PMID 28601132
- [Background] Khan BA, Perkins AJ, Gao S, Hui SL, Campbell NL, Farber MO, Chlan LL, Boustani MA. The Confusion Assessment Method for the ICU-7 Delirium Severity Scale: A Novel Delirium Severity Instrument for Use in the ICU. Crit Care Med. 2017 May;45(5):851-857. doi: 10.1097/CCM.0000000000002368. PMID 28263192
- [Background] Shenkin SD, Fox C, Godfrey M, Siddiqi N, Goodacre S, Young J, Anand A, Gray A, Hanley J, MacRaild A, Steven J, Black PL, Tieges Z, Boyd J, Stephen J, Weir CJ, MacLullich AMJ. Delirium detection in older acute medical inpatients: a multicentre prospective comparative diagnostic test accuracy study of the 4AT and the confusion assessment method. BMC Med. 2019 Jul 24;17(1):138. doi: 10.1186/s12916-019-1367-9. PMID 31337404
- [Background] Maclullich AM, Anand A, Davis DH, Jackson T, Barugh AJ, Hall RJ, Ferguson KJ, Meagher DJ, Cunningham C. New horizons in the pathogenesis, assessment and management of delirium. Age Ageing. 2013 Nov;42(6):667-74. doi: 10.1093/ageing/aft148. Epub 2013 Sep 25. PMID 24067500
- [Background] Tieges Z, Evans JJ, Neufeld KJ, MacLullich AMJ. The neuropsychology of delirium: advancing the science of delirium assessment. Int J Geriatr Psychiatry. 2018 Nov;33(11):1501-1511. doi: 10.1002/gps.4711. Epub 2017 Apr 9. PMID 28393426
- [Background] Ely EW, Margolin R, Francis J, May L, Truman B, Dittus R, Speroff T, Gautam S, Bernard GR, Inouye SK. Evaluation of delirium in critically ill patients: validation of the Confusion Assessment Method for the Intensive Care Unit (CAM-ICU). Crit Care Med. 2001 Jul;29(7):1370-9. doi: 10.1097/00003246-200107000-00012. PMID 11445689
- [Background] Kaplan PW. The EEG in metabolic encephalopathy and coma. J Clin Neurophysiol. 2004 Sep-Oct;21(5):307-18. PMID 15592005
- Available data/document: Individual Participant Data Set — https://eeg.ceribell.com — This website is password protected and the de-identified individual participant data is only available to participating research sites.